CLINICAL TRIAL: NCT04048785
Title: The Effects of Behavioral Sleep Intervention on Infant Sleep and Social-emotional Development
Brief Title: Behavioral Sleep Intervention and Infant Sleep and Social-emotional Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Sijia Gu, staff of Research Department, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCMCIRB-K2018013
Record Dates: First submitted 2019-07-31; First posted 2019-08-07 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Infant Sleep Problem
Keywords: Child health care; Behavior sleep intervention; Mental health; Social emotional development
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Infants are randomly assigned to one of two groups: Behavioral Sleep Intervention or Control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Trial participants and individuals assessing the outcomes are blinded to the participant's condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Infant sleep monitoring (Actigraphy and sleep dairy) and parental surveys
- Infant behavioral sleep intervention (Experimental): Interventionists collaborate with the family to design a tailored sleep intervention strategy, which involves appropriate sleep schedule and bedtime routine, putting the child to bed while still sleepy rather than when already asleep, and waiting 1 to 2 minutes before attending to the child during nocturnal awakenings. Parents are educated to implement the behavioral protocol at bedtime and subsequent night wakings.
  Interventions: Other: Behavioral sleep intervention

INTERVENTIONS:
Other: Behavioral sleep intervention — The intervention consists of an infant behavioral sleep protocol. In the tailored intervention approach, parents are asked to implement the behavioral protocol at bedtime and at subsequent night wakings.
  Arms: Infant behavioral sleep intervention

SUMMARY:
An estimated 30-50% of infants have frequent problematic night wakings. Sleep disturbances have been linked to various adverse outcomes in children, including social-emotional development delay. Despite some evidence of the effectiveness of Infant behavioral sleep intervention, the benefits on children's social-emotional development are worthy of further exploration. The aim of this study is to evaluate the efficacy of behavioral sleep interventions on improving infant sleep and social-emotional development. Infants with behavioral sleep disturbances are randomized into one of the two conditions: Behavioral sleep intervention or no treatment. And infant sleep and social-emotional development were assessed for both group at baseline, and four and eight weeks after sleep intervention.

DETAILED DESCRIPTION:
Study Design: The study design was a parallel group RCT with two groups (Behavioral sleep intervention and Control) and three assessment points. Sleep was assessed by actigraphy (and sleep daily) and parent-reported Brief Infant Sleep Questionnaire (BISQ) during the week before behavioral sleep intervention, four weeks and eight weeks after sleep intervention. Other measures were collected during a laboratory visit scheduled at the end of each of the three assessment.

Participants: Participants were recruited through web-based media advertisements. Approximately 100 participants will be randomized to behavioral sleep intervention condition or a control condition. Inclusion criteria were: 1) infant age range 5-18 months; 2) significant sleep problem lasting at least 2 weeks, manifested in an average of ≥30 minutes sleep onset latency, and/or ≥2 awakenings per night based on parent reports; and 3) two-parent families with both mother and father willing to participate in study procedures. Exclusion criteria were: 1) infant pervasive developmental disorder or significant medical illness; and 2) any concurrent treatment for infant sleep problems.

Study Procedure: Participants are screened via telephone. Caregivers of the intervention group were instructed to establish tailored behavioral sleep intervention strategies. Control families received no sleep intervention. For infants with sleep problems in control group, any sleep treatment in health care services should be recorded. Infant social-emotional development were assessed by Ages & Stages Questionnaires: Social-Emotional2 (ASQ:SE2) and behaviors in Still face experiment. During the experiment, the mother and infant engage in a three-step interaction: 1) playing"peek-a-boo" for 60 seconds; 2) mother maintaining a neutral facial expression while looking at the child, not smiling, talking, or touching for 120 seconds still-face (SF) episode; 3) maternal re-engagement with the infant to"peek-a-boo" for a 60 seconds reunion (RE) episode. The study was approved by the Institutional Review Board of Shanghai Children's Medical Center and all parents provided written informed consent.

Intervention: One clinical psychologist and one pediatrician delivered the intervention. The intervention was performed at Shanghai Children's Medical Center after parents signed the informed consent form. Interventionists collaborate with the family to design a tailored sleep intervention strategy, which involves appropriate sleep schedule and bedtime routine, putting the child to bed while still sleepy rather than when already asleep, caregivers should minimize their involvement after putting the infant to bed, and waiting 1 to 2 minutes before attending to the child during nocturnal awakenings. Parents are educated to implement the behavioral protocol at bedtime and subsequent night wakings. Furthermore, families of intervention group received a e-booklet describing their intervention and cell phone support weekly.

Measures: Infant sleep is assessed by Actigraphy and parent-report (sleep diary and Brief Infant Sleep Questionnaire, BISQ); Infant social-emotional development is evaluated by Ages & Stages Questionnaires: Social-Emotional2 (ASQ:SE2), and behaviors (facial expression, gaze, and self-comforting) in three separate dimensions during the Still face experiment.

ELIGIBILITY:
Inclusion Criteria:

* Infant age range 5-18 months;
* Sleep problem lasting at least 2 weeks, manifested in an average of ≥30 minutes sleep onset latency, and/or ≥2 awakenings per night based on parent reports;
* Both mother and father willing to participate in study procedures.

Exclusion Criteria:

* Infant pervasive developmental disorder or significant medical illness;
* Any concurrent treatment for infant sleep problems.

Ages: 5 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant sleep measured by Actigraphy | changes from baseline, 4 weeks and 8 weeks after the intervention
  Sleep-wake patterns are determined using actigraphy, which has been established as a valid method to objectively assess sleep in the infant's natural setting. Parents were asked to attach a actigraph (Motionlogger, Ambulatory Monitoring, Inc., Ardsley, NY, USA) to their child's ankle for 7 days at each assessment period. Data was scored using the Sadeh algorithm, which is the most commonly used analysis method in pediatric populations. Sleep diaries were completed by parents and used to identify and amend any irregularities in actigraphic data. The following actigraphic sleep metrics were used: 1) wake after sleep onset (WASO); 1) sleep of latency (SOL); and 3) number of awakenings (NW).
Infant sleep measured by Brief Infant Sleep Questionnaire | changes from baseline, 4 weeks and 8 weeks after the intervention
  The BISQ is a well-validated sleep questionnaire aimed at assessing parent-reported infant sleep patterns. Parents completed the BISQ at each assessment point. The derived measures used in this study were: (1) sleep onset latency (SOL); (2) wake after sleep onset (WASO); and (3) number of awakenings.

SECONDARY OUTCOMES:
Infant social-emotional development | changes from baseline, 4 weeks and 8 weeks after the intervention
  ASQ:SE2 consists of a set of multiple choice questions that should be completed by caregivers of the infant. The questions are divided into forms according to age, and ask about behaviour in different areas: 1) self-regulation; 2) conformity; 3) adaptive functioning; 4) autonomy; 5) affect; 6) social communication; and 7) interaction with other persons. It makes it possible to detect if there is a risk in infant social-emotional development.
  Developed as an ecologically-valid procedure for assessing emotion regulation (the foundation of the social-emotional development) in the context of parent-child interaction, the Still face procedure enables examination of infant modulation of affect, attention, and behavior in socially-stressful situations.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Fan, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Paap MC, Haraldsen IR, Breivik K, Butcher PR, Hellem FM, Stormark KM. The Link between Peer Relations, Prosocial Behavior, and ODD/ADHD Symptoms in 7-9-Year-Old Children. Psychiatry J. 2013;2013:319874. doi: 10.1155/2013/319874. Epub 2012 Dec 18. PMID 24286065
- [Background] Slomski A. Chronic mental health issues in children now loom larger than physical problems. JAMA. 2012 Jul 18;308(3):223-5. doi: 10.1001/jama.2012.6951. No abstract available. PMID 22797621
- [Background] Kahn M, Sheppes G, Sadeh A. Sleep and emotions: bidirectional links and underlying mechanisms. Int J Psychophysiol. 2013 Aug;89(2):218-28. doi: 10.1016/j.ijpsycho.2013.05.010. Epub 2013 May 24. PMID 23711996
- [Background] Baglioni C, Spiegelhalder K, Lombardo C, Riemann D. Sleep and emotions: a focus on insomnia. Sleep Med Rev. 2010 Aug;14(4):227-38. doi: 10.1016/j.smrv.2009.10.007. Epub 2010 Feb 6. PMID 20137989
- [Background] Yoo SS, Gujar N, Hu P, Jolesz FA, Walker MP. The human emotional brain without sleep--a prefrontal amygdala disconnect. Curr Biol. 2007 Oct 23;17(20):R877-8. doi: 10.1016/j.cub.2007.08.007. No abstract available. PMID 17956744
- [Background] Vandekerckhove M, Cluydts R. The emotional brain and sleep: an intimate relationship. Sleep Med Rev. 2010 Aug;14(4):219-26. doi: 10.1016/j.smrv.2010.01.002. Epub 2010 Apr 2. PMID 20363166
- [Background] Payne JD, Chambers AM, Kensinger EA. Sleep promotes lasting changes in selective memory for emotional scenes. Front Integr Neurosci. 2012 Nov 21;6:108. doi: 10.3389/fnint.2012.00108. eCollection 2012. PMID 23181013
- [Background] van der Helm E, Gujar N, Walker MP. Sleep deprivation impairs the accurate recognition of human emotions. Sleep. 2010 Mar;33(3):335-42. doi: 10.1093/sleep/33.3.335. PMID 20337191
- [Background] Zohar D, Tzischinski O, Epstein R. Effects of energy availability on immediate and delayed emotional reactions to work events. J Appl Psychol. 2003 Dec;88(6):1082-93. doi: 10.1037/0021-9010.88.6.1082. PMID 14640818
- [Background] Fernandez-Mendoza J, Vela-Bueno A, Vgontzas AN, Ramos-Platon MJ, Olavarrieta-Bernardino S, Bixler EO, De la Cruz-Troca JJ. Cognitive-emotional hyperarousal as a premorbid characteristic of individuals vulnerable to insomnia. Psychosom Med. 2010 May;72(4):397-403. doi: 10.1097/PSY.0b013e3181d75319. Epub 2010 Apr 5. PMID 20368477
- [Background] Palmer CA, Alfano CA. Sleep and emotion regulation: An organizing, integrative review. Sleep Med Rev. 2017 Feb;31:6-16. doi: 10.1016/j.smrv.2015.12.006. Epub 2016 Jan 14. PMID 26899742
- [Background] Crichton GE, Symon B. Behavioral Management of Sleep Problems in Infants Under 6 Months--What Works? J Dev Behav Pediatr. 2016 Feb-Mar;37(2):164-71. doi: 10.1097/DBP.0000000000000257. PMID 26836644
- [Background] Heckman JJ. Schools, Skills, and Synapses. Econ Inq. 2008 Jun;46(3):289. doi: 10.1111/j.1465-7295.2008.00163.x. PMID 20119503
- [Background] Weisman O, Magori-Cohen R, Louzoun Y, Eidelman AI, Feldman R. Sleep-wake transitions in premature neonates predict early development. Pediatrics. 2011 Oct;128(4):706-14. doi: 10.1542/peds.2011-0047. Epub 2011 Sep 12. PMID 21911350
- [Background] Sun W, Wang G, Jiang Y, Song Y, Dong S, Lin Q, Deng Y, Zhu Q, Jiang F. Six-month-old infant long sleepers prefer a human face. Sleep Med. 2016 Nov-Dec;27-28:28-31. doi: 10.1016/j.sleep.2016.08.018. Epub 2016 Oct 31. PMID 27938915
- [Background] Hunnius S, de Wit TC, Vrins S, von Hofsten C. Facing threat: infants' and adults' visual scanning of faces with neutral, happy, sad, angry, and fearful emotional expressions. Cogn Emot. 2011 Feb;25(2):193-205. doi: 10.1080/15298861003771189. PMID 21432667
- [Background] Korkmaz B. Theory of mind and neurodevelopmental disorders of childhood. Pediatr Res. 2011 May;69(5 Pt 2):101R-8R. doi: 10.1203/PDR.0b013e318212c177. PMID 21289541
- [Background] Alexander GM, Wilcox T, Woods R. Sex differences in infants' visual interest in toys. Arch Sex Behav. 2009 Jun;38(3):427-33. doi: 10.1007/s10508-008-9430-1. Epub 2008 Nov 19. PMID 19016318
- [Background] Wilcox T, Biondi M. fNIRS in the developmental sciences. Wiley Interdiscip Rev Cogn Sci. 2015 May-Jun;6(3):263-83. doi: 10.1002/wcs.1343. Epub 2015 Feb 23. PMID 26263229
- [Background] Hiscock H, Bayer J, Gold L, Hampton A, Ukoumunne OC, Wake M. Improving infant sleep and maternal mental health: a cluster randomised trial. Arch Dis Child. 2007 Nov;92(11):952-8. doi: 10.1136/adc.2006.099812. Epub 2006 Dec 7. PMID 17158146
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Whiteford+HA%2C+Degenhardt+L%2C+Rehm+J%2C+Baxter+AJ%2C+Ferrari+AJ%2C+Erskine+HE%2C+Charlson+FJ%2C+Norman+RE%2C+Flaxman+AD%2C+Johns+N%2C+Burstein+R%2C+Murray+CJ%2C+Vos+T.+Global+burden+of+disease+attributable+to+mental+and+substance+use+disorders%3A+findings+from+the+Global+Burden+of+Disease+Study
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Kessler+RC%2C+Berglund+P%2C+Demler+O%2C+Jin+R%2C+Merikangas+KR%2C+Walters+EE.+Lifetime+prevalence+and+age-of-onset+distributions+of+DSM-IV+disorders+in+the+National+Comorbidity+Survey+Replication.+Arch+Gen+Psychiatry%2C+2005%3B+62(6)%3A+593-602.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=The+link+between+peer+relations%2C+prosocial+behavior%2C+and+ODD%2FADHD+symptoms+in+7-+9-year-old+children
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Chronic+mental+health+issues+in+children+now+loom+larger+than+physical+problems
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Kahn+M%2C+Sheppes+G%2C+Sadeh+A.+Sleep+and+emotions%3A+bidirectional+links+and+underlying+mechanisms.+Int+J+Psychophysiol.+2013%3B89(2)
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Baglioni+C%2C+Spiegelhalder+K%2C+Lombardo+C%2C+Riemann+D.+Sleep+and+emotions%3A+a+focus+on+insomnia.+Sleep+Med+Rev.+2010%3B14(4)%3A227-23
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Yoo+SS%2C+Gujar+N%2C+Hu+P%2C+Jolesz+FA%2C+Walker+MP.+The+human+emotional+brain+without+sleep--a+prefrontal+amygdala+disconnect.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Vandekerckhove+M%2C+Cluydts+R.+The+emotional+brain+and+sleep%3A+an+intimate+relationship.+Sleep+Med+Rev.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Payne+JD%2C+Chambers+AM%2C+Kensinger+EA.+Sleep+promotes+lasting+changes+in+selective+memory+for+emotional+scenes.+Front
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=van+der+Helm+E%2C+Gujar+N%2C+Walker+MP.+Sleep+deprivation+impairs+the+accurate+recognition+of+human+emotions.+Sleep.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Zohar+D%2C+Tzischinski+O%2C+Epstein+R.+Effects+of+energy+availability+on+immediate+and+delayed+emotional+reactions+to+work+events.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Fernández-Mendoza+J%2C+Vela-Bueno+A%2C+Vgontzas+AN%2C+Ramos-Platón+MJ%2C+Olavarrieta-Bernardino+S%2C+Bixler+EO%2C+De+la+Cruz-Troca+JJ.+Cognitive-emotional+hyperarousal+as+a+premorbid+characteristic+of+individuals+vulnerable+to+insomnia.+Psychosom+Med
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=almer+CA%2C+Alfano+CA.+Sleep+and+emotion+regulation%3A+An+organizing%2C+integrative+review.+Sleep+Med+Rev.+2017
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Crichton+GE%2C+Symon+B.+Behavioral+Management+of+Sleep+Problems+in+Infants+Under+6+Months--What+Works%3F
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Heckman%2C+JJ.+Schools%2C+skills+and+synapses.+Econ+Inq%2C2008%3B46(3)%3A289.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Weisman+O%2C+Magori-Cohen+R%2C+Louzoun+Y%2C+Eidelman+AI%2C+Feldman+R.+Sleep-wake+transitions+in+premature+neonates+predict+early+development.+Pediatrics.+2011%3B128(4)%3A706-14.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Sun+W%2C+Wang+G%2C+Jiang+Y%2C+Song+Y%2C+Dong+S%2C+Lin+Q%2C+Deng+Y%2C+Zhu+Q%2C+Jiang+F.+Six-+month-old+infant+long+sleepers+prefer+a+human+face.Sleep+Med.+2016%3B27-28%3A28-3
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Hunnius+S%2C+de+Wit+TCJ%2C+Vrins+S%2C+von+Hofsten+C.+Facing+threat%3A+infants'+and+adults%27+visual+scanning+of+faces+with+neutral%2C+happy%2C+sad%2C+angry%2C+and+fearful+emotional+expressions
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Korkmaz+B.+Theory+of+mind+and+neurodevelopmental+disorders+of+childhood.+Pediatr+Res%2C+2
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Alexander+GM%2C+Wilcox+T%2C+Woods+R.+Sex+differences+in+infants'+visual+interest+in+toys.+Arch+Sex+Behav%2C
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Wilcox+T%2C+Biondi+M.+fNIRS+in+the+developmental+sciences.+Wiley+Interdiscip+Rev+Cogn+Sci.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Hiscock+H%2C+Bayer+J%2C+Gold+L%2C+Hampton+A%2C+Ukoumunne+OC%2C+Wake+M.+Improving+infant+sleep+and+maternal+mental+health%3A+a+cluster+randomised+trial.